CLINICAL TRIAL: NCT03118531
Title: Evaluation of the Clinical Safety and Efficacy of the 34/38 mm Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System in the Treatment of Suitable Subjects According to the Indication for Use.
Brief Title: China Resolute Integrity 34/38 mm Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT16003RES001
Record Dates: First submitted 2017-03-30; First posted 2017-04-18 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Heart Disease; Stenotic Coronary Lesion; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
Keywords: Long Lesion; In-stent Late Lumen Loss (LLL); Major Adverse Cardiac Events (MACE); MYOCARDIAL INFARCTION (MI); TARGET VESSEL REVASCULARIZATION (TVR); TARGET LESION REVASCULARIZATION (TLR); Target Vessel Failure (TVF); Target Lesion Failure (TLF); Stent Thrombosis (ST)
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary Stent (Experimental): Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System (34/38 mm)
  Interventions: Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System(34/38 mm)

INTERVENTIONS:
Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System(34/38 mm) — The stenting procedure should be performed according to the Instructions for Use that is provided with each 34/38 mm Resolute Integrity stent.

SUMMARY:
To evaluate the clinical safety and efficacy in Chinese subjects, eligible for percutaneous transluminal coronary angioplasty (PTCA) in lesions amenable to treatment with a 34/38 mm Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, the Instructions for Use of the Resolute Integrity 34/38 mm stent
* The subject can have either a single lesion, or two lesions located in separate target vessels treated during the index procedure. Each lesion length needs to be ≤35mm with at least one lesion length >27mm and≤ 35mm and amenable for treatment with a Resolute Integrity 34/38 mm stent

Key Exclusion Criteria:

* STEMI within 24 hours
* Left main disease
* Bifurcation disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Late lumen loss, in stent | 9 months (m)
  Late lumen loss measured by quantitative coronary angiography (QCA)

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  Defined as death, myocardial infarction (Q wave and non-Q wave), or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods
Death | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  All death
Myocardial infarction | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  All MI, and Target Vessel Myocardial Infarction (TVMI)
All revascularizations | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  Target Legion Revascularization (TLR), Target Vessel Revascularization (TVR) and Non-TVR
Target Vessel Failure (TVF) | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  TVF
Target Lesion Failure (TLF) | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  TLF
Stent Thrombosis (ST) | 30 days, 6 and 9 months, 1, 2, 3, 4, and 5 years
  ST
Device Success | At the end of index procedure, an expected average of 3 days
  The attainment of <50% residual stenosis of the target lesion using only the assigned device.
  The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using the assigned device only. These measurements will be made by the independent angiographic core laboratory.
Lesion Success | At the end of index procedure, an expected average of 3 days
  The attainment of <50% residual stenosis of the target lesion using any percutaneous method.
  The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using any percutaneous method. These measurements will be made by the independent angiographic core laboratory.
Procedure Success | Duration of hospital stay, an expected average of 5 days
  The attainment of <50% residual stenosis of the target lesion and no in-hospital MACE.
  The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using any percutaneous method without the occurrence of MACE during the hospital stay. These measurements will be made by the independent angiographic core laboratory.
In-stent and in-segment percent diameter stenosis (%DS) | 9 months
  In-stent and in-segment percent diameter stenosis (%DS)
In-stent and in-segment binary restenosis rate | 9 months
  In-stent and in-segment binary restenosis rate
In-stent and in-segment minimal luminal diameter (MLD) | 9 months
  In-stent and in-segment minimal luminal diameter (MLD)
In-segment late luminal loss | 9 months
  In-segment late luminal loss

CONTACTS AND LOCATIONS:
Overall Officials: Lianglong Chen, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian